CLINICAL TRIAL: NCT06911593
Title: Relationship of Arterial Stiffness Value With Hemodynamic Parameters in Patients Undergoing Cardiac Surgery
Brief Title: Arterial Stiffness and Hemodynamics in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mustafa Aydemir, Specialist, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 2022/3982
Record Dates: First submitted 2025-03-13; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Hypotension; Anesthesia-Induced Hypotension; Arterial Stiffness; Cardiovascular Diseases
Keywords: Arterial stiffness; Cardiac surgery; Doppler ultrasonography; Pulse wave velocity; Stiffness index
MeSH Terms: conditions — Hypotension; Cardiovascular Diseases | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: In our study, a single group was analyzed without comparisons to another group. Ultrasonographic measurements were performed within a single patient cohort.
  Interventions: Diagnostic Test: Doppler ultrasonography

INTERVENTIONS:
Diagnostic Test: Doppler ultrasonography — The delay time was determined as the time difference between the onset of the Doppler waveform and the R-wave on the electrocardiogram(ECG) of the USG device. The distance between the carotid and femoral arteries, where imaging was performed, was then measured. This distance was divided by the delay time to calculate the carotid-femoral pulse wave velocity(PWV) in meters per second, which was considered a measure of arterial stiffness.

SUMMARY:
Background:

Hypotension during the induction of anesthesia is a significant clinical condition associated with increased perioperative morbidity and mortality. This study aims to evaluate whether hypotension occurring during anesthesia induction can be predicted using arterial stiffness and stiffness index parameters measured by ultrasonography. Additionally, the study investigates potential associations between arterial stiffness parameters and intraoperative hemodynamic variables, vasoactive drug use, length of stay in the hospital and intensive care unit (ICU), and mortality.

Methods:

This prospective study was conducted in patients scheduled for elective open cardiac surgery. The predictive value of arterial stiffness, measured by ultrasonography, for identifying hypotension during anesthesia induction was assessed. Carotid-femoral pulse wave velocity (PWV) and stiffness index (β index) were used as indicators of arterial stiffness.

DETAILED DESCRIPTION:
Background:

Hypotension during anesthesia induction is a serious clinical condition that may lead to adverse perioperative outcomes such as myocardial ischemia, renal hypoperfusion, and neurological complications. In cardiac surgery, hypotension during induction can compromise myocardial perfusion and increase the risk of ischemic events. In patients with significant coronary artery disease, a sudden drop in systemic blood pressure can reduce coronary perfusion pressure, potentially resulting in left ventricular dysfunction and hemodynamic instability. Therefore, careful hemodynamic management and appropriate use of vasopressors during anesthesia induction are critical to improving perioperative outcomes in open cardiac surgery.

Arterial stiffness refers to the reduced elasticity of arterial walls due to loss of elastic tissue. It increases with age and is associated with a higher risk of cardiovascular disease. Arterial stiffness can be assessed using ultrasonography (USG) or applanation tonometry. Ultrasonographic pulse wave velocity (PWV) measurements are comparable to those obtained via tonometry. Arterial stiffness has become nearly synonymous with PWV, but research on stiffness index and ultrasonographic stiffness measurements remains limited. The predictive role of arterial stiffness in anesthesia-induced hypotension has not been adequately evaluated. This study was designed to address this gap by evaluating whether arterial stiffness and stiffness index measured by USG can predict hypotension during anesthesia induction. Exploratory analyses also examined associations with intraoperative hemodynamic changes, vasoactive drug use, ICU and hospital stay, and mortality.

Methods:

This prospective study was conducted between October 1, 2022, and May 1, 2023, at a university hospital. Ethical approval was obtained from the institutional review board. Patients scheduled for elective cardiac surgery were evaluated. Arterial stiffness and stiffness index values measured by ultrasonography, along with intraoperative and postoperative clinical data, were analyzed. Informed consent was obtained from all participants.

Participants:

Patients aged 18-85 years scheduled for elective cardiac surgery were included. Exclusion criteria included arrhythmia, end-stage renal disease, left ventricular ejection fraction <35%, reoperation, emergency surgery, body mass index >40 kg/m², and incomplete data. Upon arrival in the operating room, standard monitoring was initiated, including ECG, SpO₂, and invasive arterial pressure via radial artery cannulation under local anesthesia. All arterial stiffness measurements were performed by a single clinician after sedation with midazolam and fentanyl. Measurements were conducted in the supine position, followed by anesthesia induction and central venous catheterization. Hemodynamic parameters, hypotension episodes, and vasoactive agent use were recorded throughout the surgical procedure. After surgery, participants were transferred to the intensive care unit.

Measurements - Pulse Wave Velocity (PWV):

A 3-lead ECG was connected to the patient. Measurements were taken in the supine position with the head turned to the left. A sector probe was placed at the bifurcation of the right sternocleidomastoid muscle to visualize Doppler waveforms of the carotid artery. A linear probe was used to measure maximum and minimum diameters of the carotid artery. The femoral artery was imaged below the inguinal ligament. Doppler signals were recorded from both sites simultaneously with ECG. The time delay between the ECG R-wave and the start of the Doppler waveform was measured across three cardiac cycles and averaged. The distance between the measurement points was divided by the delay time to calculate PWV (m/s). This value represented arterial stiffness.

The stiffness index (β) was calculated using the maximum and minimum diameters of the carotid artery and systolic/diastolic blood pressure values:

β = [ln(Systolic BP / Diastolic BP)] / [(Systolic Diameter - Diastolic Diameter) / Diastolic Diameter] The vasoactive inotropic score (VIS) was used to assess the degree of vasopressor and inotropic support. A VIS ≥10 is considered an independent risk factor for increased morbidity and mortality.

Data Collection:

Baseline systolic, diastolic, and mean arterial pressures and heart rate values were recorded pre-induction, pre-intubation, and within the first 10 minutes post-intubation. Additional hemodynamic parameters such as systolic pressure variation (SPV), pulse pressure variation (PPV), and central venous pressure (CVP) were also collected. Intraoperative hypotension was defined as systolic arterial pressure (SAP) <90 mmHg. Thresholds of <80 mmHg and <70 mmHg were also explored. The types and doses of vasoactive and inotropic agents used during surgery, including during cardiopulmonary bypass, were recorded. VIS values were calculated and analyzed in relation to arterial stiffness parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 who underwent elective cardiac surgery

Exclusion Criteria:

* Arrhythmia
* End-stage renal failure on dialysis
* Left ventricular ejection fraction <35%
* Reoperation
* Emergency surgery
* Body mass index >40
* Missing data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral Pulse Wave Velocity (PWV) | Baseline (prior to anesthesia induction)
  PWV will be calculated by dividing the distance between the carotid and femoral measurement sites by the time delay between the R-wave on the ECG and the onset of the Doppler waveform. Measurements will be obtained via Doppler ultrasonography prior to anesthesia induction. The average of three consecutive cardiac cycles will be used to ensure accuracy.
  Unit of Measure:
  Meters per second (m/s)

SECONDARY OUTCOMES:
Stiffness Index (β) | Within the first 15 minutes following anesthesia induction
  The stiffness index (β) will be calculated using the following formula:
  β = [ln(Systolic BP / Diastolic BP)] / [(Systolic Diameter - Diastolic Diameter) / Diastolic Diameter] This calculation will be based on carotid artery diameters measured by ultrasound and non-invasive blood pressure measurements.
  Unit of Measure:
  Unitless ratio
Vasoactive Inotropic Score (VIS) | From anesthesia induction until the end of surgery (up to 6 hours)
  VIS will be calculated to quantify the amount of vasopressor and inotropic support administered during surgery. The formula is as follows:
  VIS = Dopamine (mcg/kg/min) + Dobutamine (mcg/kg/min) + 100 × Epinephrine (mcg/kg/min) + 100 × Norepinephrine (mcg/kg/min) + 10 × Milrinone (mcg/kg/min) + 10,000 × Vasopressin (units/kg/min)
  Unit of Measure:
  Numeric score
Length of Stay in the Intensive Care Unit (ICU) | From admission to the ICU until discharge from the ICU (up to 14 days)
  The number of days each participant spends in the intensive care unit (ICU) following surgery will be recorded. This outcome will be used to explore potential associations with arterial stiffness parameters.
  Unit of Measure:
  Days
Length of Stay in the Hospital | From the day of surgery until hospital discharge (up to 30 days)
  The total number of days each participant remains hospitalized after surgery will be recorded. This exploratory outcome will be analyzed in relation to arterial stiffness and stiffness index values.
  Unit of Measure:
  Days

CONTACTS AND LOCATIONS:
Locations (1):
- NecmettinEU, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Mustafa Aydemir Medical Doctor, Necmettin Erbakan University, Medical School, Department of Anesthesiology and Reanimation, Konya, Turkey drmustafaaydemir02@gmail.com ORCID: orcid.org/0000-0002-6289-7031